CLINICAL TRIAL: NCT04906538
Title: Objective Results of Anterior Cruciate Ligament Reconstruction With and Without Internal Suture Augmentation Technique
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed abdelaziz Ramadan, orthopedic surgery registrar, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 310 2018
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Rolimeter; ACLR; internal suture augmentation; IKDC score; Lysholm score
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anterior cruciate ligament reconstruction with internal suture augmentation technique (Active Comparator): This group will be operated by using all-inside ACLR technique with internal suture augmentation technique
  Interventions: Procedure: all- inside anterior cruciate ligament reconstruction
- anterior cruciate ligament reconstruction without internal suture augmentation technique (Active Comparator): This group will be operated by using all-inside ACLR technique without internal suture augmentation technique
  Interventions: Procedure: all- inside anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: all- inside anterior cruciate ligament reconstruction — all- inside anterior cruciate ligament reconstruction with internal suture augmentation technique

SUMMARY:
The purpose of this study is (1) To report, compare and corelate the patient reported outcomes (PRO) (IKDC score, Lysholm Score) and range of motion (ROM) among patients following hamstring autograft ACLR with and without independent suture tape reinforcement against objective laxity test using Lachmeter. (2) Rate of complications and reoperation.

DETAILED DESCRIPTION:
Investigators performed a randomized control trial in two groups utilizing All- inside ACLR. Group I was augmented by suture tape and Group 2 without suture tape augmentation. From October 2018 to June 2020, 20 patients underwent all-inside ACL reconstruction with internal suture augmentation technique (Group I, Brace group) and the other 18 patients underwent all- inside ACL reconstruction without internal suture augmentation technique (Group II, non-brace group). Demographic data (age, sex, side of injury, time since injury), manual assessment (Lachman test, pivot shift test, ROM), PROs (IKDC score, Lysholm score) and Lachmeter examination were collected and analyzed at fixed time points during follow-up period as mean duration of follow up in our series was 18 months ± 3.4 (range, 12-24 months).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 years old.
* Patients will be diagnosed as ACL tear by the following:

I. History of knee traumatic event. II. Clinical examination (ant. Drawer test, Lachman test and pivot shift test). III. Radiological evidence of ACL tear by MRI.

Exclusion Criteria:

* Other intra or extra articular knee injuries.
* Previous ACL surgery on the affected knee.
* Bilateral ACL injuries.
* Significant Articular surface injury.
* Medical comorbidities
* Patients with malalignment (genu varum. Genu valgum and Genu recurvatum)
* Neuromuscular disorders

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Lachmeter examination | 9 months
  objective measurement of knee laxity
Lysholm score | 9 months
  subjective knee functional score (0 - 100) score. 100 is better in function
International Knee Documentation score (IKDC) score | 9 months
  subjective knee functional score (0 - 100) score. 100 is better in function

SECONDARY OUTCOMES:
knee ROM | 9 months
  post- operative knee ROM

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Khater, MD, Principal Investigator — Professor of orthopedic surgery
Locations (1):
- Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
study protocol and abstract

REFERENCES:
- [Background] Sobhy MH, Khater AH, Hassan MR, El Shazly O. Do functional outcomes and cuff integrity correlate after single- versus double-row rotator cuff repair? A systematic review and meta-analysis study. Eur J Orthop Surg Traumatol. 2018 May;28(4):593-605. doi: 10.1007/s00590-018-2145-7. Epub 2018 Feb 13. PMID 29442181